CLINICAL TRIAL: NCT00602745
Title: A Multicenter, Open-Label, Randomized Study Comparing Efficacy and Safety of S-1 as Single Agent Versus 5-FU Bolus for the Treatment of Patients With Metastatic Pancreatic Cancer Previously Treated With a Gemcitabine-Based Regimen
Brief Title: S-1 Versus 5-FU Bolus in Metastatic Pancreatic Cancer Patients Previously Treated With Gemcitabine-Based Regimen
Acronym: S-1 Pancreas
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Following the termination of development and commercialization agreement for S-1 with Taiho Pharmaceutical
Sponsor: Sanofi (Industry)
Collaborators: Taiho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EFC10203; S-1 - FI
Record Dates: First submitted 2008-01-16; First posted 2008-01-28 (Estimated); Last update posted 2016-05-26 (Estimated); Status verified 2016-04

CONDITIONS: Pancreatic Neoplasm; Neoplasm Metastasis
Keywords: pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasm Metastasis | interventions — S 1 (combination); Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 5-Fluorouracil (Active Comparator)
  Interventions: Drug: 5-Fluorouracil
- S-1 (Experimental)
  Interventions: Drug: S-1

INTERVENTIONS:
Drug: S-1 — oral administration
  Arms: S-1
Drug: 5-Fluorouracil — intravenous bolus
  Arms: 5-Fluorouracil

SUMMARY:
The primary objective of this study is to determine whether S-1 increases overall survival when compared to 5-Fluorouracil (5-FU) in patients with metastatic pancreatic cancer previously treated with a gemcitabine-based therapy.

The secondary objectives are to compare: progression free survival, overall response rate, clinical benefit and improvement in tumor related symptoms and also to assess overall safety and pharmacokinetics of S-1.

ELIGIBILITY:
Inclusion Criteria:

* Cytologically or histologically confirmed evidence of adenocarcinoma of the exocrine pancreas
* Metastatic disease previously treated with a gemcitabine-based regimen

Exclusion Criteria:

* Locally advanced disease
* More than one prior chemotherapy-line for advanced pancreatic disease
* Prior treatment with fluoropyrimidines for advanced pancreatic cancer
* Eastern Cooperative Oncology Group (ECOG) performance status >or= 2
* Poor kidney, liver or bone marrow functions
* Any serious active disease or co-morbid condition, which in the opinion of the principle investigator, will interfere with the safety or with compliance with the study
* Unable to swallow capsules
* Hypersensitivity history to any of the constituents of the study medications or fluoropyrimidines
* Concurrent participation in another clinical trial or treatment with any other anticancer therapy

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2008-02; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Overall Survival | study period

SECONDARY OUTCOMES:
Progression Free Survival | every 6 weeks
Overall Response Rate according to RECIST criteria | every 6 weeks
Clinical Benefit assessed by Time to Symptoms Worsening (TTSW) | every 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (17):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, Vienna, Austria
- Sanofi-Aventis Administrative Office, São Paulo, Brazil
- Sanofi-Aventis Administrative Office, Laval, Canada
- Sanofi-Aventis Administrative Office, San José, Costa Rica
- Sanofi-Aventis Administrative Office, Hørsholm, Denmark
- Sanofi-Aventis Administrative Office, Paris, France
- Sanofi-Aventis Administrative Office, Athens, Greece
- Sanofi-Aventis Administrative Office, Mixco, Guatemala
- Sanofi-Aventis Administrative Office, Budapest, Hungary
- Sanofi-Aventis Administrative Office, Netanya, Israel
- Sanofi-Aventis Administrative Office, Ocean Business Plaza, Panama
- Sanofi-Aventis Administrative Office, Lima, Peru
- Sanofi-Aventis Administrative Office, Bucharest, Romania
- Sanofi-Aventis Administrative Office, Midrand, South Africa
- Sanofi-Aventis Administrative Office, Bromma, Sweden
- Sanofi-Aventis Administrative Office, Mégrine, Tunisia